CLINICAL TRIAL: NCT01940588
Title: Neuropsychoanalytic Treatment of Failed Back Surgery Syndrome-Opioid Dependence
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: University at Buffalo (Other)
Responsible Party: Sponsor
Other Study IDs: 1 - bjohnson
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Neuropsychoanalytic treatment: Outpatient detoxification, intensive neuropsychoanalytic therapy, low dose naltrexone, monthly evaluations for six months - case series approach.
  Interventions: Behavioral: Neuropsychoanalytic therapy

INTERVENTIONS:
Behavioral: Neuropsychoanalytic therapy — Psychotherapy, medication management

SUMMARY:
Opioid Dependent Patients who have failed back surgery syndrome are detoxified and treated with a neuropsychoanalytic paradigm.

DETAILED DESCRIPTION:
Patients were detoxified from opioid analgesics and treated with NSAIDs and other non-opioid analgesics, received neuropsychoanalytic therapy and low dose naltrexone. Patients kept a daily diary of: 0 - 10 pain, 0 - 10 function, hours worked, amount of alcohol drunk, illicit and licit drug use, number of health care provider appointments attended, number of self-help groups meetings attended across each of the six months of study. Six month outcomes of this approach with primary outcomes being sobriety, pain scores and function scores.

ELIGIBILITY:
Inclusion Criteria:

1. Have failed back surgery syndrome.
2. Have evidence of Opioid Dependence by meeting DSM-IV criteria and by Drug Abuse Screening Test > 4. (In case of a difference in these two measures, clinical staff will talk with the patient to adjudicate the difference.)
3. Over 18
4. Be able to understand spoken and written English
5. Reside within 30 miles of the site of treatment for ease of followup
6. Have health insurance or other ability to pay for treatment

Exclusion Criteria:

1. Homeless
2. Unable to give consent (e.g. neurological disorders, dementia, psychosis)
3. Co-occurring incapacitating psychiatric disorder such as schizophrenia
4. Pregnant
5. Financial incentive to stay ill, such as a pending disability claim
6. Member of a vulnerable population, including prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with failed back surgery syndrome and opioid use disorder 18 years of age and older
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Improvement of pain | Six months
  Detoxified patients followed for whether their pain improved.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Johnson, M.D., Principal Investigator — State University of New York - Upstate Medical University